CLINICAL TRIAL: NCT06549920
Title: Danish Breast Cancer Group Internal Mammary Node Study
Acronym: DBCG IMN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, Professor, Danish Breast Cancer Cooperative Group
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG IMN protocol
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Internal mammary node irradiation; Node-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal mammary node irradiation (Experimental): Patients with right-sided breast cancer tumors were allocated to internal mammary node irradiation.
  Interventions: Radiation: Internal mammary node irradiation
- No internal mammary node irradiation (No Intervention): Patients with left-sided breast cancer tumors were allocated to no internal mammary node irradiation.

INTERVENTIONS:
Radiation: Internal mammary node irradiation — Irradiation of the internal mammary nodes in intercostal space 1-4.
  Other Names: IMNI
  Arms: Internal mammary node irradiation

SUMMARY:
The DBCG IMN study is a nationwide prospective population-based cohort study allocating node-positive breast cancer patients with right-sided tumors to internal mammary node irradiation (IMNI) and patients with left-sided tumors to no IMNI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macrometastatic node-positive breast cancer treated with loco-regional radiotherapy.

Exclusion Criteria:

* Prior malignancies, bilateral breast cancer, neoadjuvant systemic therapy, recurrence before radiotherapy, and non-standard radiotherapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7630 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2034-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 15-years.
  Censored at end of study or by emigration.

SECONDARY OUTCOMES:
Breast cancer mortality | 15-years.
  Censored at end of study or by emigration.
Distant recurrences | 15-years.
  Censored at end of study or by emigration. Death by any cause was regarded as competing event.

IPD SHARING:
Plan to Share IPD: Yes
Data may be requested at the DBCG RT committee and the DBCG board.
Time Frame: Undecided.
Access Criteria: DBCG board.

REFERENCES:
- [Derived] Nielsen AWM, Thorsen LBJ, Ozcan D, Matthiessen LW, Maae E, Milo MLH, Nielsen MH, Tramm T, Overgaard J, Offersen BV; DBCG RT Committee. Internal mammary node irradiation in 4541 node-positive breast cancer patients treated with newer systemic therapies and 3D-based radiotherapy (DBCG IMN2): a prospective, nationwide, population-based cohort study. Lancet Reg Health Eur. 2024 Dec 12;49:101160. doi: 10.1016/j.lanepe.2024.101160. eCollection 2025 Feb. PMID 39810969